CLINICAL TRIAL: NCT06974565
Title: An Open-label, Randomized, Cross-over, Single Dose Study in Healthy Participants to Assess the Pharmacokinetics of AZD2389 When Administered Alone and in Combination With Quinidine
Brief Title: A Study to Investigate the Pharmacokinetics of AZD2389 in Healthy Participants When Administered Alone and in Combination With Quinidine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D7930C00006
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Advanced Chronic Liver Disease; Healthy Participants
Keywords: Hepatic Fibrosis; Fibroblast Activation Protein Inhibitor
MeSH Terms: conditions — Liver Cirrhosis | interventions — Quinidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Experimental): Participants will receive a single dose of Treatment A (AZD2389) in Period 1 and a single dose of Treatment B (AZD2389 + quinidine) in Period 2.
  Interventions: Drug: AZD2389; Drug: Quinidine
- Sequence BA (Experimental): Participants will receive a single dose of Treatment B (AZD2389 + quinidine) in Period 1 and a single dose of Treatment A (AZD2389) in Period 2.
  Interventions: Drug: AZD2389; Drug: Quinidine

INTERVENTIONS:
Drug: AZD2389 — AZD2389 will be administered orally.
Drug: Quinidine — Quinidine will be administered orally.

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) and safety of AZD2389 when administered alone and in combination with quinidine in healthy participants.

DETAILED DESCRIPTION:
This is a 2-way cross-over study to evaluate the effect of quinidine on the PK of AZD2389.

The study will include 2 Treatments - Treatment A - AZD2389 Treatment B - AZD2389 + quinidine

The study will comprise -

1. A Screening Period of maximum 28 days.
2. Period 1: single dose administration of Treatment A or Treatment B on Day 1. Period 2 will start after a washout period of at least 7 days.
3. Period 2: single dose of alternate treatment on Day 8.
4. A Follow-up Visit: participants will return for a Follow-up Visit, 7 to 14 days after the last AZD2389 PK sample in Period 2.

Participants will be randomized to one of the 2 treatment sequences -

1. Sequence AB: Treatment A in Period 1, Treatment B in Period 2.
2. Sequence BA: Treatment B in Period 1, Treatment A in Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential) participants with suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of non-childbearing potential must be confirmed at the Screening Visit.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the study specific contraception methods from the time of first administration of study intervention administration until 3 months after the study Follow-up Visit.
* Have a body mass index between 18 and 32 kg/m2, inclusive, and weigh at least 50 kg at the Screening Visit.

Exclusion Criteria:

* History of any clinically important disease or disorder.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important abnormalities in hematology, clinical chemistry, urinalysis, coagulation results or other laboratory values and vital signs.
* Any positive result on Screening for serum hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV).
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead electrocardiogram (ECG) at Screening.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Current smokers or those who have smoked or used nicotine products within the previous 3 months prior to screening.
* Positive screen for drugs of abuse, or alcohol or cotinine at Screening.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* History of hypersensitivity to dipeptidyl peptidase 4 (DPP4) inhibitors.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Ratio of Test treatment (AZD2389 + quinidine) to Reference treatment (AZD2389) based on maximum observed plasma concentration (RCmax) | Day 1 to Day 10
  To assess the effect of quinidine on the PK of AZD2389.
Ratio of Test treatment (AZD2389 + quinidine) to Reference treatment (AZD2389) based on area under concentration-time curve from time 0 to infinity (RAUCinf) | Day 1 to Day 10
  To assess the effect of quinidine on the PK of AZD2389.
Ratio of Test treatment (AZD2389 + quinidine) to Reference treatment (AZD2389) based on area under concentration-time curve from time 0 to the last quantifiable concentration (RAUClast) | Day 1 to Day 10
  To assess the effect of quinidine on the PK of AZD2389.

SECONDARY OUTCOMES:
Apparent total body clearance (CL/F) of AZD2389 | Day 1 to Day 10
  To assess the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Volume of distribution (apparent) following extravascular administration (based on terminal phase) (Vz/F) of AZD2389 | Day 1 to Day 10
  To assess the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Terminal elimination half-life (t1/2λz) of AZD2389 | Day 1 to Day 10
  To assess the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Time to reach maximum observed concentration (tmax) of AZD2389 | Day 1 to Day 10
  To assess the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Maximum observed plasma concentration (Cmax) of AZD2389 | Day 1 to Day 10
  To assess the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) of AZD2389 | Day 1 to Day 10
  To assess the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Area under concentration-time curve from time zero to infinity (AUCinf) of AZD2389 | Day 1 to Day 10
  To assess the plasma PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Renal Clearance (CLR) of AZD2389 from plasma | Day 1 to Day 10
  To assess the urine PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 (fe[t1-t2]) of AZD2389 | Day 1 to Day 10
  To assess the urine PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Individual and cumulative amount of unchanged drug excreted into urine from time t1 to time t2 (Ae[t1-t2]) of AZD2389 | Day 1 to Day 10
  To assess the urine PK of AZD2389 when AZD2389 is administered alone or in combination with quinidine.
Percent change from baseline in fibroblast activation protein (FAP) inhibition | Baseline, Day 1 to Day 10
  To assess the pharmacodynamics (PD) of AZD2389 by assessment of inhibition of FAP activity in plasma after single oral dose of AZD2389 alone or in combination with quinidine.
Number of participants with Adverse Events (AEs) | From Screening (Day -28 to Day -2) to Follow-up visit (upto 8 weeks)
  To assess the safety and tolerability of a single oral dose of AZD2389 alone or in combination with quinidine in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/